CLINICAL TRIAL: NCT03104153
Title: Effect of Early Removal of Wound Drains After Mastectomy or Lymph Node Dissection on Clinical Outcome and Quality of Life in Breast Cancer Patients
Brief Title: Effect of Early Removal of Wound Drains After Mastectomy or Lymph Node Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S58129
Record Dates: First submitted 2017-03-27; First posted 2017-04-07 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2017-03

CONDITIONS: Draining Wound; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Output-based (No Intervention)
- Early-removal (Active Comparator)
  Interventions: Procedure: Early-drain removal

INTERVENTIONS:
Procedure: Early-drain removal — Drain removal at hospital discharge
  Arms: Early-removal

SUMMARY:
To compare early drain removal versus output-based drain removal, assessing the following end-points:

Clinical : risk of seroma and infection, woundhealing, duration of wound care and drain output versus volume of seroma.

Quality of life : drain-induced pain, discomfort due to seroma or drain, sleep disturbance and implications on daily activities.

Cost-effectiveness

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for breast cancer surgery with placement of suction drainage
* Female or male
* Age > 18 years
* All stages of disease (inclusion is independent of TNM-classification)

Exclusion Criteria:

* Patients scheduled for breast cancer surgery without placement of suction drains
* No informed consent: Patient refuses participation OR is not able to give a written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 3 weeks
  Improve the quality of life, wich will be measured by a questionnaire with some specific questions.

IPD SHARING:
Plan to Share IPD: No